CLINICAL TRIAL: NCT00886262
Title: Low Dose Vasopressin for Renal Protection During Liver Transplantation
Brief Title: Study to Evaluate if the Drug Vasopressin Protects the Kidneys for Patients Undergoing Liver Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vasopressin HR #17345
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-08

CONDITIONS: Liver Failure
Keywords: liver transplantation; vasopressin; renal function; hypotension; creatinine; urine output; diuretics; vasopressors; hemodynamic stability
MeSH Terms: conditions — Liver Failure; Diabetes Insipidus; Hypotension | interventions — Vasopressins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vasopressin (Experimental)
  Interventions: Drug: Vasopressin
- Normal saline placebo (Placebo Comparator)
  Interventions: Drug: Normal saline placebo

INTERVENTIONS:
Drug: Vasopressin — Patients randomly assigned to the experimental arm of the study will receive vasopressin 0.5U/hr IV (20 U vasopressin in 250mL of 0.9% NaCL to infuse at a rate of 6.25mL/hr) via internal jugular catheter. Vasopressin infusion is started at the time of incision and is stopped at the time abdominal closure is completed
  Arms: Vasopressin
Drug: Normal saline placebo — Patients randomly assigned to the placebo arm of the study will receive placebo (0.9% NaCl to infuse at a rate of 6.25 mL/hr) via internal jugular catheter
  Arms: Normal saline placebo

SUMMARY:
The purpose of this study is evaluate the medication vasopressin for its ability to preserve kidney function in patients undergoing liver transplantation.

DETAILED DESCRIPTION:
Renal failure is a common complication of liver disease. Hepatorenal syndrome is caused by a dysfunctional global circulation in the setting of liver disease: Increased flow to the mesenteric circulation is a contributor to decreased blood flow to the kidneys (1). Renal failure often worsens in the perioperative period of liver transplantation since the kidneys are further stressed by reduced flow due to inferior venacava occlusion, decreased blood flow to the kidneys from anesthetics, as well as hypotension from volume shifts, such as when large volumes of ascites are removed. Renal failure is a cause of major morbidity and mortality in patients undergoing liver transplantation.

Vasopressin is a logical choice of therapy in this context as the effects of the drug work to particularly increase renal blood flow and glomerular filtration rate due to the location of specific vasopressin receptors within the renal vasculature. It has been suggested that the use of splanchnic (and systemic) vasoconstrictors such as terlipressin (a vasopressin analog) or alpha-1-adrenoceptor agonists (midodrine or noradrenaline) may improve renal function in patients with type 1 Hepatorenal Syndrome.

Six studies (with only one randomized study in a small series of patients) have shown that terlipressin improves renal function in these patients (2-7). This drug is available in Europe, but not in the United States. However, while anesthesiologists commonly use vasopressin during liver transplantation in the setting of hepatorenal syndrome or vasodilatory shock, the validity of this practice for its effects on renal function and outcomes has not been rigorously studied (8-10). Therefore, the purpose of this study is to evaluate the effects of low-dose vasopressin on intraoperative and perioperative renal function in liver transplant patients.

This study will be a randomized, double-blind controlled trial performed in adult liver transplant patients coming to surgery for chronic liver disease; the major end-points of analyses are renal function tests in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* undergoing liver transplant
* ability to provide informed consent. If patient is unable to give informed consent i.e. hepatic encephalopathy, consent may be obtained from the patient's legally authorized representative

Exclusion Criteria:

* < 18 years of age
* renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D McEvoy, MD, Principal Investigator — Medical University of South Carolina; Scott T Reeves, MD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Moreau R, Lebrec D. The use of vasoconstrictors in patients with cirrhosis: type 1 HRS and beyond. Hepatology. 2006 Mar;43(3):385-94. doi: 10.1002/hep.21094. PMID 16496352
- [Background] Uriz J, Gines P, Cardenas A, Sort P, Jimenez W, Salmeron JM, Bataller R, Mas A, Navasa M, Arroyo V, Rodes J. Terlipressin plus albumin infusion: an effective and safe therapy of hepatorenal syndrome. J Hepatol. 2000 Jul;33(1):43-8. doi: 10.1016/s0168-8278(00)80158-0. PMID 10905585
- [Background] Mulkay JP, Louis H, Donckier V, Bourgeois N, Adler M, Deviere J, Le Moine O. Long-term terlipressin administration improves renal function in cirrhotic patients with type 1 hepatorenal syndrome: a pilot study. Acta Gastroenterol Belg. 2001 Jan-Mar;64(1):15-9. PMID 11322061
- [Background] Moreau R, Durand F, Poynard T, Duhamel C, Cervoni JP, Ichai P, Abergel A, Halimi C, Pauwels M, Bronowicki JP, Giostra E, Fleurot C, Gurnot D, Nouel O, Renard P, Rivoal M, Blanc P, Coumaros D, Ducloux S, Levy S, Pariente A, Perarnau JM, Roche J, Scribe-Outtas M, Valla D, Bernard B, Samuel D, Butel J, Hadengue A, Platek A, Lebrec D, Cadranel JF. Terlipressin in patients with cirrhosis and type 1 hepatorenal syndrome: a retrospective multicenter study. Gastroenterology. 2002 Apr;122(4):923-30. doi: 10.1053/gast.2002.32364. PMID 11910344
- [Background] Halimi C, Bonnard P, Bernard B, Mathurin P, Mofredj A, di Martino V, Demontis R, Henry-Biabaud E, Fievet P, Opolon P, Poynard T, Cadranel JF. Effect of terlipressin (Glypressin) on hepatorenal syndrome in cirrhotic patients: results of a multicentre pilot study. Eur J Gastroenterol Hepatol. 2002 Feb;14(2):153-8. doi: 10.1097/00042737-200202000-00009. PMID 11981339
- [Background] Ortega R, Gines P, Uriz J, Cardenas A, Calahorra B, De Las Heras D, Guevara M, Bataller R, Jimenez W, Arroyo V, Rodes J. Terlipressin therapy with and without albumin for patients with hepatorenal syndrome: results of a prospective, nonrandomized study. Hepatology. 2002 Oct;36(4 Pt 1):941-8. doi: 10.1053/jhep.2002.35819. PMID 12297842
- [Background] Solanki P, Chawla A, Garg R, Gupta R, Jain M, Sarin SK. Beneficial effects of terlipressin in hepatorenal syndrome: a prospective, randomized placebo-controlled clinical trial. J Gastroenterol Hepatol. 2003 Feb;18(2):152-6. doi: 10.1046/j.1440-1746.2003.02934.x. PMID 12542598
- [Background] Csete M. IARS 2007 Review Course Lectures: Anesthesia for Liver Transplantation. Anes Analg 2007; 104:19-24,2007.
- [Background] Roth JV. The use of vasopressin bolus to treat refractory hypotension secondary to reperfusion during orthotopic liver transplantation. Anesth Analg. 2006 Jul;103(1):261. doi: 10.1213/01.ANE.0000215232.42488.6D. No abstract available. PMID 16790680
- [Background] De Wolf AM. Preoperative optimization of patients with liver disease. Curr Opin Anaesthesiol. 2005 Jun;18(3):325-31. doi: 10.1097/01.aco.0000169242.03754.cc. PMID 16534358

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vasopressin | Normal Saline Placebo
Started | 8 | 10
Completed | 8 | 7
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vasopressin | Normal Saline Placebo | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 58 [36 to 68] | 55.1 [30 to 69] | 56.4 [30 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Creatinine Levels
Time Frame: baseline to 48 hours postop
Measure: Mean (Full Range); unit: MG/DL
Arm/Group | Vasopressin | Normal Saline Placebo
Number analyzed (Participants) | 8 | 10
MG/DL | 0.5 [0.1 to 0.8] | 0.55 [0.1 to 1.3]

2. Primary Outcome: Change in Urine Output
Time Frame: 24 hours to 48 hours postop
Measure: Mean (Full Range); unit: mL
Arm/Group | Vasopressin | Normal Saline Placebo
Number analyzed (Participants) | 8 | 10
mL | 1353 [160 to 2830] | 731 [10 to 1550]

3. Secondary Outcome: Count of Participants Who Needed Diuretics Postoperatively
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Vasopressin | Normal Saline Placebo
Number analyzed (Participants) | 8 | 10
Participants | 4 | 1

4. Secondary Outcome: Count of Patient Who Need Vasopressers in the Perioperative Period
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Vasopressin | Normal Saline Placebo
Number analyzed (Participants) | 8 | 10
Participants | 3 | 4

ADVERSE EVENTS:
Arm/Group | Vasopressin | Normal Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes